CLINICAL TRIAL: NCT00651209
Title: A Single-arm, Multinational, Two Year Study Evaluating the Efficacy and Safety of lead-in Telbivudine for 24 Weeks With or Without Tenofovir Treatment Intensification in Adult Patients With HBeAg-positive Chronic Hepatitis B.
Brief Title: A Single-arm Study Evaluating the Efficacy and Safety of Telbivudine With or Without add-on Tenofovir in Adults With HBeAg-positive Chronic Hepatitis B (CHB)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600A2410
Record Dates: First submitted 2008-03-18; First posted 2008-04-02 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, chronic; Telbivudine; Tenofovir; Roadmap Concept
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir; Telbivudine

ARMS (1):
- 1 (Experimental): Sub-group 1- continue telbivudine if HBV DNA non-detectable at week 24 Sub-group 2- tenofovir added to telbivudine in patients if HBV DNA detectable at week 24
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Tenofovir — All patients receive 600 mg/day, oral telbivudine for 24 weeks. Patients with non-detectable HBV DNA continue 600 mg/day, oral telbivudine for the remaining treatment period (Sub-group 1) Patients with detectable HBV DNA receive 300 mg/day, oral tenofovir plus 600 mg/day, oral telbivudine for the remaining treatment period (Sub-group 2)
  Other Names: Sebivo; Tyzeka; Viread

SUMMARY:
This study will evaluate the use of telbivudine for patients with HBeAg-positive CHB with an option to intensify treatment at Week 24 by adding tenofovir for patients who do not achieve HBV DNA non-detectability.

ELIGIBILITY:
Inclusion criteria

* Male or female, at least 18 years of age.
* Documented HBeAg positive CHB defined by all of the following:
* Clinical history compatible with CHB
* Detectable serum HBsAg at the Screening visit and at least 6 months prior
* HBeAg positive at the Screening visit
* HBeAb negative at the Screening visit
* Serum HBV DNA level ≥ 5 log10 copies/mL, as determined by the COBAS Amplicor HBV PCR assay (LLOD = 300 copies / mL) at the central study laboratory at Screening visit
* Evidence of chronic liver inflammation, documented by previous history of elevated serum ALT and /or AST levels (at least two elevated ALT or AST values spanning six months or more, documented in available records) with or without prior liver biopsy that is consistent with CHB
* For patients with cirrhosis, clinical history compatible with compensated liver disease
* Elevated serum ALT level (1.3 - 10 x ULN) at the Screening visit
* Patient is willing and able to comply with the study drug regimen and all other study requirements.
* The patient is willing and able to provide written informed consent to participate in the study.

Exclusion criteria

* Patients will be excluded from the study for any of the following:
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures.
* Patient is pregnant or breastfeeding.
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means. The exception of the aforementioned criteria will be given if they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/ml (IU/L) or 6 weeks post surgical bilateral oophorectomy with or without hysterectomy or have been surgically sterilized (e.g., bilateral tubal ligation) or the patient must agree to use two methods of birth control. This is any combination of hormonal contraception (implantable, patch, oral or injection), IUD, male or female condom with spermicidal gel, diaphragm, sponge or cervical cap. Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-HCG) during Screening.
* Is a male who is capable of reproduction, defined as all men physiologically capable of producing sperm,including men whose career, lifestyle, or sexual orientation precludes intercourse with a female partner and men who have been sterilized (vasectomy) or whose partners have been sterilized by surgical bilateral oophorectomy with or without hysterectomy, bilateral tubal ligation or other means, UNLESS the female partner meets the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/ml (IU/L) or the patient must agree to use two methods of birth control. This is any combination of hormonal contraception (implantable, patch ,oral or injection), IUD, male or female condom with spermicidal gel, diaphragm, sponge or cervical cap.
* Patient is co-infected with HCV, HDV, or HIV.
* Patients who have previously been involved in a trial with telbivudine.
* Patient has received nucleoside or nucleotide drugs whether approved or investigational at any time.
* Patient has received IFN or other immunomodulatory treatment in the 12 months before Screening for this study.
* Patient has a history of or clinical signs/symptoms of hepatic decompensation such as ascites, esophageal variceal bleeding, hepatic encephalopathy, hepatorenal syndrome, hepatic hydrothorax, hepatopulmonary syndrome or spontaneous bacterial peritonitis.
* Patient has a medical condition that requires prolonged or frequent use of systemic acyclovir or famciclovir.
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
* Patients with previous findings suggestive of possible HCC, should have the disease ruled out prior to entrance into the study.
* Patient has one or more additional known primary or secondary causes of liver disease, other than CHB, including steatohepatitis and autoimmune hepatitis among other liver diseases. Note: Gilbert's syndrome and Dubin-Johnson syndrome are not considered exclusion criteria for this study.
* History of any other acute or chronic medical condition that in the opinion of the investigator would make the patient unsuitable for inclusion into the study.
* Patient is currently abusing alcohol or illicit drugs, or has a history of alcohol abuse or illicit substance abuse within the preceding two years. Please refer to Appendix 3.
* Patient has a medical condition that requires frequent or prolonged use of systemic corticosteroids, although topical and inhaled corticosteroids are allowed.
* Patient has a history of clinical and laboratory evidence of chronic renal insufficiency defined as an estimated serum creatinine clearance < 50 mL/min using the Cockcroft-Gault method.
* Patient has a medical condition requiring the chronic or prolonged use of potentially hepatotoxic drugs or nephrotoxic drugs.
* Patient has any other concurrent medical or social condition likely to preclude compliance with the schedule of evaluations in the protocol, or likely to confound the efficacy or safety observations of the study.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* Patient has a history of myopathy, myositis, or persistent muscle weakness.
* Patient has any of the following laboratory values during Screening:

Hemoglobin <11 g/dL (110 g/L) for men or <10 g/dL (100 g/L) for women Total WBC <3,500/mm3 (3.5 x 109/Liter) Absolute neutrophil count (ANC) <1,500/mm3 (1.5 x 109/Liter) Platelet count <75,000/mm3 (75 x 109/Liter) Serum amylases or lipase ≥ 1.5 x ULN Serum albumin <3.3 g/dL (33g/L) Total bilirubin ≥ 2.0 mg/dL (34.2 µmol/L) Estimated calculated serum creatinine clearance < 50 mL/min ( 0.48 ml/s) using the Cockcroft-Gault method with lean or ideal body weight; see Glossary of Terms (Cockcroft 1976) AFP > 50 ng/mL or µg/L (requires further work up per local medical standards)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-02; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to determine if telbivudine early non-responders can achieve an antiviral response with the addition of tenofovir. | at week 52

SECONDARY OUTCOMES:
To estimate the rate of virologic breakthrough up to week 48 and week 104 To assess the rate of treatment-emergent genotypically confirmed HBV resistance associated with viral breakthrough up to weeks 48 and 104 and 104 | at week 52 and 104

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (4):
- Novartis, Buenos Aires, Argentina
- Novartis, São Paulo, Brazil
- Novartis, Frankfurt, Germany
- Novartis, Bangkok, Thailand

REFERENCES:
- [Derived] Piratvisuth T, Komolmit P, Tanwandee T, Sukeepaisarnjaroen W, Chan HL, Pessoa MG, Fassio E, Ono SK, Bessone F, Daruich J, Zeuzem S, Cheinquer H, Pathan R, Dong Y, Trylesinski A. 52-week efficacy and safety of telbivudine with conditional tenofovir intensification at week 24 in HBeAg-positive chronic hepatitis B. PLoS One. 2013;8(2):e54279. doi: 10.1371/journal.pone.0054279. Epub 2013 Feb 4. PMID 23390496